CLINICAL TRIAL: NCT00380575
Title: A 4-Day, Double-Blind, Placebo-Controlled, Multicenter Study of IV YM087 (CI-1025) to Assess Efficacy and Safety in Patients With Euvolemic or Hypervolemic Hyponatremia
Brief Title: Study of IV YM087 to Assess Efficacy and Safety in Patients With Euvolemic or Hypervolemic Hyponatremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 087-CL-027
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Hyponatremia
Keywords: hyponatremia; hypervolemic; euvolemic; vasopressins; YM087
MeSH Terms: conditions — Hyponatremia; Diabetes Insipidus | interventions — conivaptan

INTERVENTIONS:
Drug: YM087

SUMMARY:
This study will investigate the application of a vasopressin antagonist in the treatment of hyponatremia most likely caused by inappropriate AVP secretion. The population studied will include patients with euvolemic or hypervolemic hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* Serum sodium levels 115 to < 130mEq/L
* Euvolemic or Hypervolemic hyponatremia

Exclusion Criteria:

* Clinical evidence of volume depletion or dehydration
* Untreated severe hypothyroidism, hyperthyroidism, or adrenal insufficiency
* Uncontrolled brady-or tachyarrhythmias requiring pacemaker placement or treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2000-08; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome will be change from baseline in serum sodium over the duration of treatment. The primary safety outcome will be safety parameters (e.g., adverse events, vital signs, EGG, laboratory measurements).

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (47):
- United States (27):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tuscon, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Santa Rosa, California
  - Miami, Florida
  - Plantation, Florida
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Shreveport, Louisiana
  - Worchester, Massachusetts
  - Petoskey, Michigan
  - Minneapolis, Minnesota
  - Rolla, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - New York, New York
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Columbia, South Carolina
  - Sioux Falls, South Dakota
  - Chattanooga, Tennessee
  - Norfolk, Virginia
  - Salem, Virginia
  - Huntington, West Virginia
  - Madison, Wisconsin
- Canada (2):
  - Drummondville, Quebec
  - Montreal 2 Sites, Quebec
- Israel (9):
  - Ashkelon
  - Beersheba
  - Haifa 2 Sites
  - Holon
  - Jerusalem
  - Rehovot
  - Safed
  - Tel Aviv
  - Tel Litwinsky
- South Africa (9):
  - Bloemfontein
  - Buff
  - Durban
  - East London
  - eManzimtoti
  - Johannesburg
  - Lyttelton Manor
  - Port Elizabeth
  - Pretoria

REFERENCES:
- [Background] Zeltser D, Rosansky S, van Rensburg H, Verbalis JG, Smith N; Conivaptan Study Group. Assessment of the efficacy and safety of intravenous conivaptan in euvolemic and hypervolemic hyponatremia. Am J Nephrol. 2007;27(5):447-57. doi: 10.1159/000106456. Epub 2007 Jul 26. PMID 17664863
- [Background] Verbalis JG, Zeltser D, Smith N, Barve A, Andoh M. Assessment of the efficacy and safety of intravenous conivaptan in patients with euvolaemic hyponatraemia: subgroup analysis of a randomized, controlled study. Clin Endocrinol (Oxf). 2008 Jul;69(1):159-68. doi: 10.1111/j.1365-2265.2007.03149.x. Epub 2008 Jul 1. PMID 18034777